CLINICAL TRIAL: NCT02048852
Title: Manipulating Tobacco Constituents in Female Menthol Smokers
Acronym: Menthol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H14-120-1; 1R01DA036486-01 (NIH)
Record Dates: First submitted 2014-01-27; First posted 2014-01-29 (Estimated); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Nicotine Dependence
Keywords: menthol; nicotine
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Reduced Nicotine Content -Non Menthol (Experimental): Switch from own brand of cigarette to SPECTRUM research cigarettes (NRC 200-Reduced Nicotine Content cigarette) which contain 0.07mg nicotine yield without menthol.
  Interventions: Other: Reduced Nicotine Content- Non Menthol
- Reduced Nicotine Content- Menthol (Experimental): Switch from own brand of cigarette to Reduced Nicotine Research Cigarettes which contain 0.07mg nicotine yield with Menthol
  Interventions: Other: Reduced Nicotine Content- Menthol
- Conventional Nicotine Content- Menthol (Active Comparator): Allow own brand of Conventional Nicotine-Menthol Cigarette. No research cigarettes used.
  Interventions: Other: Conventional Nicotine Content- Menthol
- Conventional Nicotine Content- Non Menthol (Experimental): Switch from own brand of cigarette to SPECTRUM research cigarette (NRC-600 Conventional Nicotine )which contains conventional nicotine yield.
  Interventions: Other: Conventional Nicotine Content- Non Menthol

INTERVENTIONS:
Other: Reduced Nicotine Content- Non Menthol — Switch from own brand of cigarette to a research cigarette with a Reduced Nicotine Content of 0.07mg nicotine yield without menthol.
  Other Names: SPECTRUM Research Cigarette - NRC 200
  Arms: Reduced Nicotine Content -Non Menthol
Other: Reduced Nicotine Content- Menthol — Switch from own brand of cigarette to Reduced nicotine level of each research cigarette to 0.07mg nicotine yield with Menthol
  Other Names: SPECTRUM Research Cigarette - RNC 201
  Arms: Reduced Nicotine Content- Menthol
Other: Conventional Nicotine Content- Menthol — Allow own brand of Conventional Nicotine-Menthol Cigarette
  Other Names: Own brand of Conventional Nicotine-Menthol Cigarette
  Arms: Conventional Nicotine Content- Menthol
Other: Conventional Nicotine Content- Non Menthol — Switch from own cigarette to a research cigarette which contains Conventional Nicotine yield.
  Other Names: SPECTRUM Research Cigarette - NRC 600
  Arms: Conventional Nicotine Content- Non Menthol

SUMMARY:
This study examines the potential effect of reducing nicotine content or menthol or both in women of reproductive age, a vulnerable population identified by the FDA in need of further research.

DETAILED DESCRIPTION:
Study is designed to address the following questions that have been outlined by the FDA as particular areas of interest:

1. What are the factors, including menthol and other flavorings that influence the appeal of tobacco products to vulnerable populations: What is the impact of these factors on cessation, switching tobacco products and multiple use?
2. What is the potential impact of modifying nicotine levels on dependence, and smoking rate and cessation, as well as patterns of switching products and use of multiple tobacco products?
3. Beyond nicotine, what other constituents enhance addictive properties?

ELIGIBILITY:
Inclusion criteria are:

1. smoking at least 5 menthol cigarettes daily for the last year;
2. able to speak, read and understand English
3. female age 18 -45 years of age;
4. stable residence;
5. not intending to quit smoking within the next 6 weeks.

Exclusion criteria are:

1. unstable psychiatric disorder (Psychiatric symptoms reported by patient or identified in medical record that cause current significant impairment in functioning or judgment such that the person's ability to come consistently for study appointments or render a decision regarding informed consent is in question.);
2. substance use which exceeds any of the following: marijuana use 3x/week, consuming 21 drinks/week or illicit drug use 1x/week;
3. history of cardiovascular disease;
4. current blood clot in arms or legs;
5. blood pressure >160/100;
6. unstable medical problems which may include but are not limited to immune system disorders, severe respiratory diseases, kidney or liver diseases, thyroid problems, substance abuse or dependence that would limit patients ability to follow experimental protocol (based on history and drug and alcohol questionaires) or other heart conditions. The study physician will determine whether a given medical condition is unstable and the appropriateness of study participation for a particular subject;
7. Serious quit attempts in the last 3 months (to ensure stability of smoking);
8. regular use (e.g., greater than weekly) of tobacco products other than cigarettes;
9. Currently using nicotine replacement or other tobacco cessation products (to minimize confounding effects of another product);
10. Pregnant or breastfeeding those planning to become pregnant,and those who are of childbearing potential and are not using an "acceptable form" of birthcontrol such as Depo-provera, Norplant, tubal ligation and barrier methods such as condoms or diaphragm.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 381 (Actual)
Dates: Start 2014-07; Primary Completion 2020-03 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
The goal of the cigarette conditions is to find the impact of varying nicotine and menthol concentrations on smoking rate and abstinence. | 12 weeks
  Alter the nicotine and menthol concentrations of cigarettes administered to subjects as randomized.

SECONDARY OUTCOMES:
Toxicant Exposure | 12 weeks
  Examine the effects of reduced nicotine and menthol removal on toxicant exposure for the outcomes-- cotinine, exhaled carbon monoxide, and urine carcinogens and other tobacco specific nitrosamines.

OTHER OUTCOMES:
Cigarette content manipulations effect on a model mediating usage | 12 Weeks
  Examine cigarette content manipulation (nicotine reduction and menthol removal) as independent variables and the number of cigarettes recorded daily as dependent variable..Measures that will be tested for include subscales of the cigarette evaluations as well as craving, affect and mood, and self-confidence
Effect of taster status | 12 Weeks
  To explore the moderating effects of supertasters with menthol assignments to predict compliance with treatment, cigarette taste and aversion. A logistic model will be used to predict post-treatment abstinence. The interaction between supertaster and menthol will test for the moderating effect.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl A Oncken, MD MPH, Principal Investigator — UCONN Health Center
Locations (2):
- United States (2):
  - UCONN Health Center, Farmington, Connecticut
  - Hartford Hospital, Hartford, Connecticut

IPD SHARING:
Plan to Share IPD: No